CLINICAL TRIAL: NCT06173791
Title: Demineralized Bone Allograft Fibers Versus Particulate In Sinus Augmentation: A Double Arm Randomized Control And Histomorphometric Study
Brief Title: Demineralized Bone Allograft Fibers Versus Particulate In Sinus Augmentation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Angela Palaiologou-Gallis, DDS, MS, Professor and Program Director, Graduate Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20230387H
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Bone Loss in Jaw
Keywords: Tooth loss; Bone Resorption; Xenograft; Allograft
MeSH Terms: conditions — Tooth Loss; Bone Resorption

STUDY DESIGN:
Intervention Model Description: This is a two-independent arm, parallel-design randomized, prospective trial designed to compare two standard of care techniques
Who Masked: Participant
Masking Description: Only investigators will know which material was used for the sinus lift.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DFDBA Fibers with DBBM (Active Comparator): After standard of care elevation of the Schneiderian membrane, a mix of DFDBA fibers with DBBM (50%-50%) will be introduced in the space created between the Schneiderian membrane and the alveolar crest of the maxilla.
  Interventions: Device: DFDBA fibers; Device: DBBM
- DFDBA Particles with DBBM (Other): After standard of care elevation of the Schneiderian membrane, a mix of DFDBA particles with DBBM (50%-50%) will be introduced in the space created between the Schneiderian membrane and the alveolar crest of the maxilla.
  Interventions: Device: DFDBA particles; Device: DBBM

INTERVENTIONS:
Device: DFDBA fibers — Bone Allograft fibers used in dental sinus reconstruction surgery
  Other Names: Demineralized Freeze Dried Bone Allograft Fibers
  Arms: DFDBA Fibers with DBBM
Device: DFDBA particles — Bone Allograft particles used in dental sinus reconstruction surgery
  Other Names: Demineralized Freeze Dried Bone Allograft Particles
  Arms: DFDBA Particles with DBBM
Device: DBBM — DBBM is routinely used in sinus augmentation to support dental implant placement and restoration of missing teeth.
  Other Names: Deproteinized Bovine Bone Mineral

SUMMARY:
The purpose of this clinical trial is to assess if the addition of DFDBA fibers to DBBM results in greater vital bone formation than the addition of DFDBA particles to DBBM.

The study team will examine the effects of the addition of DFDBA fibers to DBBM on vital bone formation. Specifically, we will assess histologically the percent vital bone formation with each of the groups during implant placement, six months after the sinus augmentation procedure. We will also evaluate the radiographic volume achieved with both groups of materials.

DETAILED DESCRIPTION:
This entire protocol involves procedures that are standard care and will randomize subjects to of one two routine care procedures. Patients needing maxillary sinus augmentation will be enrolled. There will be two subject groups in this study both of which will randomized to one of two standard care procedures. No risk or benefit is expected from being assigned to either group as both procedures are both standard care. In both groups a bone sample (core) will be obtained as a by-product of implant placement. Bone will not be extracted solely for research purposes, the bone sample attained for research will only be from bone left over after the SOC implant placement.

Allocation of subjects into test group or control group will be based on numbers drawn from a stack of sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age 18 and 89
* Patients needing sinus augmentation to support implant placement in the posterior maxilla
* Patients must be nonsmokers, former smokers, or current smokers who smoke <10 cigarettes per day, by self-report
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non- pregnant women of child-bearing potential.

Exclusion Criteria:

* Patients who disclose that they will not be able to cooperate with the follow-up schedule.
* Patients who are mentally incompetent, prisoners, or pregnant (as obtained via chart review or self-report)
* Pregnant women or women intending to become pregnant during study period
* Smokers who smoke > 10 cigarettes per day

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Vital Bone Formation | Baseline to 6 months
  Each side of the maxillary sinus will be used as a separate unit of analysis. The assumption is that each patient will have only one side of the maxillary sinus; however, it is common for some patients to need both maxillary sinuses augmented (2 sites in a single patient). Change in vital bone formation will be measured from baseline (surgery) to 6 months post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Palaiologou-Gallis, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified Individual Participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published or otherwise made available